CLINICAL TRIAL: NCT03732391
Title: A Phase II Study of Pembrolizumab Plus Carboplatin in BRCA-related Metastatic Breast Cancer
Brief Title: Phase 2 Study of Pembrolizumab+Carboplatin in Breast Related Cancer Antigens-related Metastatic Breast Cancer (PEMBRACA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: CORTESI LAURA (Other)
Responsible Party: Sponsor-Investigator, CORTESI LAURA, Principal Investigator, Azienda Ospedaliero-Universitaria di Modena
Organization: Azienda Ospedaliero-Universitaria di Modena (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PEMBRACA
Record Dates: First submitted 2018-10-31; First posted 2018-11-06 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pembrolizumab; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- single arm (Experimental): Carboplatin AUC6 EV will be given every 3 weeks in combination with Pembrolizumab 200 mg EV every 3 weeks for 6 cycles. Afterwards, the Pembrolizumab will come continued with the same schedule until unacceptable toxicity or disease progression
  Interventions: Drug: Pembrolizumab 25 MG(milligram)/ML

INTERVENTIONS:
Drug: Pembrolizumab 25 MG(milligram)/ML — Carboplatin AUC6 EV will be given every 3 weeks in combination with Pembrolizumab 200 mg EV every 3 weeks for 6 cycles. Afterwards, the Pembrolizumab will be continued with the same schedule until unacceptable toxicity or disease progression
  Other Names: Carboplatin

SUMMARY:
This is a prospective two-stage single arm phase II study to be conducted in conformance with Good Clinical Practices.

This study will enrol 53 patients, based on a two steps Simon's design.

Patients will entry into the study if the following conditions will be satisfied:

* BRCA1/2 germline mutations.
* Metastatic disease with measurable lesions will be evaluated by computed tomography or by PET (Positron Emission Tomography) scan.
* Patients must have received anthracycline and taxanes before entry into the study.

Patients will be treated with Carboplatin AUC6 (Area Under The Curve) EV (endovenous) every 3 weeks in combination with Pembrolizumab 200 mg EV every 3 weeks for 6 cycles. Afterwards, the Pembrolizumab will recontinued with the same schedule until unacceptable toxicity or disease progression.

The primary endpoint will be Objective Responses Rate (ORR) (complete answers + partial answers) evaluated according to the RECIST criteria.

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent/assent for the trial.
2. Be 18 years of age on day of signing informed consent.
3. Patients must have metastatic confirmed breast cancer
4. Disease progression by radiological techniques within 12 months prior to signing informed consent
5. Documented mutation in BRCA1 or BRCA2 genes that is predicted to be deleterious or suspected deleterious (unknown significance variants)
6. Have measurable disease based on RECIST 1.1.
7. Prior chemotherapy with anthracyclines and taxanes has to be administered in neoadjuvant or adjuvant setting.
8. Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 1. Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen
9. Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale.
10. Life expectancy of greater than 3 months
11. Demonstrate adequate organ function. All screening labs should be performed within 10 days of treatment initiation.
12. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
13. Female subjects of childbearing potential must be willing to use an adequate method of contraception as outlined in Section 5.111.2 - Contraception, for the course of the study through 120 days after the last dose of study medication.

    Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
14. Male subjects of childbearing potential must agree to use an adequate method of contraception as outlined in Section 5.11.2- Contraception, starting with the first dose of study therapy through 120 days after the last dose of study therapy.

Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
2. Has a benign variant of BRCA1/2 genes
3. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment.
4. Has a known history of active Bacillus Tuberculosis
5. Hypersensitivity to pembrolizumab or any of its excipients.
6. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
7. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
8. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
9. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
10. Has active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
11. Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
12. Has an active infection requiring systemic therapy.
13. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
14. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
15. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
16. Has received prior therapy with an anti-PD-1 (anti-programmed cell Death-1), anti-PD-L1, or anti-PD-L2 agent.
17. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
18. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV (Hepatitis C Virus) RNA [qualitative] is detected).
19. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed.

    -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2018-12-12 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
The ORR | through study completion, an average of 1 year
  objective response rate (complete response plus partial response) will be evaluated according to RECIST criteria

SECONDARY OUTCOMES:
TTP (time to tumor progression) | through study completion, an average of 1 year
  (time to tumor progression)

CONTACTS AND LOCATIONS:
Locations (1):
- AOU Modena, Modena, Italy

IPD SHARING:
Plan to Share IPD: No